CLINICAL TRIAL: NCT02753231
Title: Effects of an Exercise Program on Hepatic Metabolism and Cardiovascular Health in Overweight/Obese Adolescent From Bogota, Colombia (HEPAFIT Study)
Brief Title: Exercise Training and Hepatic Metabolism in Overweight/Obese Adolescent
Acronym: HEPAFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad de Santiago de Chile (Other); Universidad de Granada (Other); Universidad Pública de Navarra (Other); Emory University (Other); University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Robinson Ramírez-Vélez, Principal Investigator, Centro de Estudios en Medición de la Actividad Física (CEMA), Universidad Santo Tomas
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: UR-21042016
Record Dates: First submitted 2016-04-21; First posted 2016-04-27 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Obesity; Metabolic Syndrome X; Lipid Metabolism Disorders; Body Composition, Beneficial; Mental Health Wellness 1
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Lipid Metabolism Disorders; Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low physical activity program (Experimental): Three Physical Education sessions / week
  Interventions: Behavioral: Low physical activity program
- High physical activity program (Experimental): Three Physical Education sessions / week (increased volume)
  Interventions: Behavioral: High physical activity program
- Low and High physical activity program (Experimental): Three Physical Education sessions / week (increased volume and intensity)
  Interventions: Behavioral: Low and High physical activity program
- Conventional physical activity program (Active Comparator): One Physical Education sessions / week
  Interventions: Behavioral: Conventional physical activity program

INTERVENTIONS:
Behavioral: Low physical activity program — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: Low physical activity program
Behavioral: High physical activity program — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: High physical activity program
Behavioral: Low and High physical activity program — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: Low and High physical activity program
Behavioral: Conventional physical activity program — One Physical Education sessions / week
  Arms: Conventional physical activity program

SUMMARY:
The HEPAFIT Study aims to examine whether a 6-months physical education program has benefits on hepatic metabolism and cardiovascular health as well as on selected physical fitness and mental health outcomes among adolescent overweight/obese from Bogota, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity status
* 11-17 years old
* Written informed consent
* Interested in improving health and fitness

Exclusion Criteria:

* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.
* Clinical diagnosis of diabetes
* Pregnancy
* Drugs/alcohol abuse

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in hepatic fat measured by controlled attenuation parameter values (FibroScan®) | Baseline and 6 months
  Changes in hepatic fat fraction measured by controlled attenuation parameter after the 6 months intervention program

SECONDARY OUTCOMES:
Changes in liver enzymes | Baseline and 6 months
  Changes in total alanine transaminase (ALT) after the 6 months intervention program
Changes in serum lipid profile | Baseline and 6 months
  Changes in cholesterol total, LDL cholesterol, HDL cholesterol and triglycerides after the 6 months intervention program
Changes in Insulin sensitivity measured by homeostasis model assessment (HOMA) | Baseline and 6 months
  Changes in insulin sensitivity measured by homeostasis model assessment (HOMA) after the 6 months intervention program
Change from Baseline in Aerobic fitness measured on a maximum effort test | Baseline and 6 months
  Change from Baseline in Cardiorespiratory fitness measured on a maximum effort test
Change from Baseline in Muscular Fitness assessed using handgrip test (maximum handgrip strength assessment) | Baseline and 6 months
  Muscular fitness will be assessed using handgrip test (maximum handgrip strength assessment) using a standard adjustable handle analogue handgrip dynamometer T-18 TKK SMEDLY III®
Change from Baseline in Body composition | Baseline and 6 months
  Fat mass as measured by Dual Energy X-ray Absorptiometry
Changes in physical activity using accelerometry | Baseline and 6 months
  Changes in physical activity estimated by accelerometry after the 6 months intervention program
Change from Baseline in Quality & satisfaction with life by SF Community - short-form survey (SF-12™) Colombian version | Baseline and 6 months
Changes in blood pressure | Baseline and 6 months
  Changes in blood pressure after the 6 months intervention program
Changes in liver enzymes | Baseline and 6 months
  Changes in total gamma-GT after the 6 months intervention program
Changes in liver enzymes | Baseline and 6 months
  Changes in total aspartate transaminase (AST) after the 6 months intervention program
Changes in inflammatory markers after the 6 months intervention program | Baseline and 6 months
  Changes in TNF-alpha after the 6 months intervention program
Changes in inflammatory markers after the 6 months intervention program | Baseline and 6 months
  Changes in IL-6 and IL-10 after the 6 months intervention program
Changes in inflammatory markers after the 6 months intervention program | Baseline and 6 months
  Changes in C-reactive protein (CRP) after the 6 months intervention program
Change from Baseline in Body composition | Baseline and 6 months
  Lean body mass as measured by Dual Energy X-ray Absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Robinson Ramirez Velez, Ph.D, Study Chair — Universidad del Rosario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Velez R, Garcia-Hermoso A, Correa-Rodriguez M, Fernandez-Irigoyen J, Palomino-Echeverria S, Santamaria E, Correa-Bautista JE, Gonzalez-Ruiz K, Izquierdo M. Effects of Different Doses of Exercise on Inflammation Markers Among Adolescents With Overweight/Obesity: HEPAFIT Study. J Clin Endocrinol Metab. 2022 May 17;107(6):e2619-e2627. doi: 10.1210/clinem/dgac021. PMID 35038337
- [Derived] Gonzalez-Ruiz K, Correa-Bautista JE, Izquierdo M, Garcia-Hermoso A, Martinez-Vizcaino V, Lobelo F, Gonzalez-Jimenez E, Schmidt-RioValle J, Correa-Rodriguez M, Fernandez-Irigoyen J, Palomino-Echeverria S, Santamaria E, Ramirez-Velez R. Exercise dose on hepatic fat and cardiovascular health in adolescents with excess of adiposity. Pediatr Obes. 2022 Apr;17(4):e12869. doi: 10.1111/ijpo.12869. Epub 2021 Nov 4. PMID 34734674
- [Derived] Gonzalez-Ruiz K, Correa-Bautista JE, Izquierdo M, Garcia-Hermoso A, Dominguez-Sanchez MA, Bustos-Cruz RH, Garcia-Prieto JC, Martinez-Vizcaino V, Lobelo F, Gonzalez-Jimenez E, Prieto-Benavides DH, Tordecilla-Sanders A, Schmidt-RioValle J, Perez G, Ramirez-Velez R. Effects of an exercise program on hepatic metabolism, hepatic fat, and cardiovascular health in overweight/obese adolescents from Bogota, Colombia (the HEPAFIT study): study protocol for a randomized controlled trial. Trials. 2018 Jun 25;19(1):330. doi: 10.1186/s13063-018-2721-5. PMID 29941024